CLINICAL TRIAL: NCT01181024
Title: A Single Ascending Dose Tolerability and Pharmacokinetic Study of RO5303253 With a Pilot Food-effect Investigation in Healthy Subjects and Exploratory Pharmacokinetic, Pharmacodynamic, and Safety Assessments in Chronic Hepatitis C Genotype 1 Patients Following 5 Days of Oral Administration
Brief Title: A Study on Safety, Tolerability and Pharmacokinetics of RO5303253 in Healthy Volunteers and Patients With Chronic Hepatitis C Genotype 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: PP25195; 2009-018183-96
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic, Healthy Volunteer
MeSH Terms: conditions — Hepatitis C; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- A: HV ascending dose (Experimental)
  Interventions: Drug: Placebo; Drug: RO5303253
- B: HV food effect (Experimental)
  Interventions: Drug: Placebo; Drug: RO5303253
- C: Hepatitis C (Experimental)
  Interventions: Drug: Placebo; Drug: RO5303253

INTERVENTIONS:
Drug: Placebo — matching RO5303253 placebo, administered as single dose (Parts A + B) or multiple dose (Part C)
Drug: RO5303253 — Cohorts receiving single ascending doses
  Arms: A: HV ascending dose
Drug: RO5303253 — Single dose
  Arms: B: HV food effect
Drug: RO5303253 — Multiple doses
  Arms: C: Hepatitis C

SUMMARY:
This randomized, double-blind, placebo controlled, 3 part study will assess the safety, tolerability and pharmacokinetics of RO5303253 in healthy volunteers and patients with chronic hepatitis C genotype 1. In Part A, cohorts of healthy volunteers will be randomized to receive single ascending doses of RO5303253 or placebo. In Part 2, healthy volunteers will receive a single dose of RO5303253 or placebo in a cross-over design (with a washout period of at least 7 days) to assess food effects on pharmacokinetics. In Part 3, patients with chronic hepatitis C will be randomized ro receive either RO5303253 or placebo for 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers or patients with chronic hepatitis C genotype 1, 18 to 60 years of age
* Patients must be treatment-naïve for antiviral therapy for chronic hepatitis C with interferon based therapy
* Body mass index (BMI) 18 - 32 kg/m2 inclusive, minimum weight 45 kg
* Females must be surgically sterile or menopausal
* Male subjects and their partners of childbearing potential must use 2 methods of contraception throughout the study and for 70 days after the last dose

Exclusion Criteria:

* Pregnant or lactating women and male partners of women who are pregnant or lactating
* Women with reproductive potential
* Positive for hepatitis B or HIV (or hepatitis C for healthy volunteers) at screening
* For hepatitis C patients: decompensated liver disease or impaired liver function, evidence of cirrhosis documented at any time, presence or history of non-hepatitis C chronic liver disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Adverse events, laboratory parameters, ECG, blood pressure | approximately 6 months
Pharmacokinetics: Plasma and urine concentrations of RO5303253 and its main metabolite RO1080713 | approximately 6 months

SECONDARY OUTCOMES:
Effect of food intake on pharmacokinetics in healthy volunteers | Days 1-4
Pharmacodynamics (viral responses) and drug resistance profiling in chronic hepatitis C patients | From baseline to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Grafton, New Zealand